CLINICAL TRIAL: NCT02498821
Title: Time and Motion Related to PICC Insertion Process and Catheter Tip Confirmation: A Comparison Between Standard of Care (Chest X-ray) and Sherlock 3CG® TCS
Brief Title: Time and Motion Related to PICC Insertion Process and Catheter Tip Confirmation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Collaborators: KJT Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BAS-14-004
Record Dates: First submitted 2015-07-01; First posted 2015-07-15 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Indication for PICC Placement
Keywords: PICC; central catheter; vascular access
MeSH Terms: interventions — Diagnostic Imaging; Catheterization, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Chest X-ray) (Other): Correct placement of the Peripherally Inserted Central Catheter (PICC) will be confirmed using standard of care (Chest X-ray).
  Interventions: Device: Chest X-ray; Procedure: Peripherally Inserted Central Catheter (PICC)
- Sherlock 3CG® TCS (Other): Correct placement of the Peripherally Inserted Central Catheter (PICC) will be confirmed using Sherlock 3CG® TCS magnetic tracking PICC placement and ECG-based tip confirmation.
  Interventions: Device: Sherlock 3CG® TCS; Procedure: Peripherally Inserted Central Catheter (PICC)

INTERVENTIONS:
Device: Chest X-ray — A Chest X-ray will be taken after healthcare providers have inserted the PICC to make sure it is in the correct location. The X-ray can tell your healthcare providers where the PICC is and whether is has been inserted correctly.
  Arms: Standard of Care (Chest X-ray)
Device: Sherlock 3CG® TCS — The Sherlock 3CG® TCS is a device that is placed on the subject during the PICC insertion procedure, which helps your healthcare providers know where the PICC is as the healthcare providers are inserting it. It uses magnets and measures electrical activity of the heart to determine the location of the catheter in your body.
  Arms: Sherlock 3CG® TCS
Procedure: Peripherally Inserted Central Catheter (PICC) — A peripherally inserted central catheter (PICC) is a form of intravenous access that can be used for a prolonged period of time (e.g., for chemotherapy, antibiotics, total parenteral nutrition)

SUMMARY:
The purpose of the study is to evaluate differences in the time and costs between Sherlock 3CG® TCS and Chest X-ray to confirm the location of a Peripherally Inserted Central Catheter (PICC).

DETAILED DESCRIPTION:
The study is a cross-sectional, observational design, characterized as a time and motion study. The study will observe subjects and specific outcomes from the time a PICC insertion procedure begins until the subject is cleared for administration of their prescribed therapy. It will compare two approaches for PICC line placement and confirmation of PICC tip placement.

The two methods for placing and confirming PICC lines to be examined in this study are: 1) Standard of Care, defined as PICC line placement with Chest X-ray tip confirmation, and 2) Sherlock 3CG® TCS magnetic tracking PICC placement and ECG-based tip confirmation. These two approaches are currently in use, and are not investigational.

The study will evaluate the time elapsed from the beginning of PICC line placement procedure through the catheter tip confirmation (subject released for IV therapy). A researcher will observe from the time the catheter kit is opened until your catheter is cleared for administration of treatment. Limited subject follow-up includes review of subject medical records related to the PICC line placement. Subjects will be followed only up to the point at which the PICC line tip has been confirmed and the subject has been released to receive IV therapy. For most subjects, all study data will be collected on Day 1.

The study is expected to include 120 subjects, 60 subjects will have confirmed PICC line placement using Chest X-ray, and 60 will have confirmed PICC line placement using Sherlock 3CG® TCS. Each group of subjects will be from two clinical sites using either tip confirmation method, for a total of 4 study sites.

ELIGIBILITY:
Inclusion Criteria:

* Indicated for a PICC based on institutional practices.
* Able to read and comprehend English and has signed the Informed Consent Form to participate in the study.
* PICC line is placed while a study observer is available and on the study site at the time of the placement.

Exclusion Criteria:

* Infection, bacteremia, or septicemia is known or suspected.
* Body size is insufficient to accommodate the size of the implanted device.
* Known or is suspected to be allergic to materials contained in the device. Materials in the device include polyurethane, stainless steel, polyimide, silicone, polytetrafluorine (PTFE), and nickle titanium.
* Past irradiation of prospective insertion site.
* Previous episodes of venous thrombosis or vascular surgical procedures at the prospective placement site.
* Local tissue factors will prevent proper device stabilization and/or access.
* Under the age of 22.
* Receiving the PICC as a replacement with an over-the-wire exchange.
* Pregnant or lactating.
* Anatomical irregularities (structural and vascular of the central venous system) which may compromise catheter insertion in both the primary arm and contralateral arm.
* Previously enrolled in this clinical study or is participating in another clinical study that is contraindicative to the treatment or outcomes of this investigation.
* Artificial heart or heart transplant.
* Anatomical abnormalities of the central venous system.
* Atrial fibrillation or other atrial arrhythmia's in which a P wave was not consistently present on ECG.
* Clinician is unable to obtain accurate external measurement due to anatomical abnormalities or personal/medical equipment.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Tomaszewski, PhD, Principal Investigator — KJT Group, Inc.
Locations (4):
- United States (4):
  - Florida Hospital, Maitland, Florida
  - University of Maryland - Baltimore, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Unity Hospital, Rochester, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Site healthcare providers identified potential subjects referred for placement of a PICC as part of their routine care. Subjects met all eligibility criteria listed in the study protocol. Recruitment occurred between May 2015 and May 2016.
Pre-assignment Details: Three patients in the Standard of Care (Chest X-ray) arm and five patients in the Sherlock 3CG TCS arm were excluded from the study as screen failures following enrollment.
Groups:
- Standard of Care (Chest X-ray): Correct placement of the Peripherally Inserted Central Catheter (PICC) will be confirmed using standard of care (Chest X-ray).
  X-ray: A Chest X-ray will be taken after healthcare providers have inserted the PICC to make sure it is in the correct location. The X-ray can tell your healthcare providers where the PICC is and whether is has been inserted correctly.
  Peripherally Inserted Central Catheter (PICC): A peripherally inserted central catheter (PICC) is a form of intravenous access that can be used for a prolonged period of time (e.g., for chemotherapy, antibiotics, total parenteral nutrition)
- Sherlock 3CG® TCS: Correct placement of the Peripherally Inserted Central Catheter (PICC)will be confirmed using Sherlock 3CG® Tip Confirmation System (TCS) magnetic tracking PICC placement and ECG-based tip confirmation.
  Sherlock 3CG® TCS: The Sherlock 3CG® TCS is a device that is placed on the subject during the PICC insertion procedure, which helps your healthcare providers know where the PICC is as the healthcare providers are inserting it. It uses magnets and measures electrical activity of the heart to determine the location of the catheter in your body.
  Peripherally Inserted Central Catheter (PICC): A peripherally inserted central catheter (PICC) is a form of intravenous access that can be used for a prolonged period of time (e.g., for chemotherapy, antibiotics, total parenteral nutrition)
Period: Overall Study
Arm/Group | Standard of Care (Chest X-ray) | Sherlock 3CG® TCS
Started | 63 | 65
Completed | 60 | 60
Not Completed | 3 | 5
Not completed — Screen failure | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Sherlock 3CG® TCS: Correct placement of the Peripherally Inserted Central Catheter (PICC)will be confirmed using Sherlock 3CG® TCS magnetic tracking PICC placement and ECG-based tip confirmation.
  Sherlock 3CG® TCS: The Sherlock 3CG® TCS is a device that is placed on the subject during the PICC insertion procedure, which helps your healthcare providers know where the PICC is as the healthcare providers are inserting it. It uses magnets and measures electrical activity of the heart to determine the location of the catheter in your body.
  Peripherally Inserted Central Catheter (PICC): A peripherally inserted central catheter (PICC) is a form of intravenous access that can be used for a prolonged period of time (e.g., for chemotherapy, antibiotics, total parenteral nutrition)
- Total: Total of all reporting groups
Arm/Group | Standard of Care (Chest X-ray) | Sherlock 3CG® TCS | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Full Range); unit: years] | 56.22 [23 to 88] | 61.75 [25 to 93] | 58.985 [23 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 29 | 51
  Male | 38 | 31 | 69
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120
Urgency of PICC Order [Count of Participants; unit: Participants]
  Very urgent (STAT) | 0 | 0 | 0
  Greater urgency than normal | 23 | 6 | 29
  Not urgent | 37 | 54 | 91

OUTCOME MEASURES:

1. Primary Outcome: Time From Initiation of Procedure (Opening of PICC Kit) to Catheter Tip Confirmation (Release for IV Therapy).
Time Frame: Usually ranges from 0 to 300 minutes from initiation of procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Standard of Care (Chest X-ray) | Sherlock 3CG® TCS
Number analyzed (Participants) | 60 | 60
minutes | 176.32 (249.84) | 33.93 (25.63)

2. Secondary Outcome: Total Number of Chest X-rays Performed Per Subject
Time Frame: Measured from initiation to completion of procedure (usually from 0 to 300 minutes)
Measure: Mean (Full Range); unit: Chest X-rays
Arm/Group | Standard of Care (Chest X-ray) | Sherlock 3CG® TCS
Number analyzed (Participants) | 60 | 60
Chest X-rays | 1.25 [0 to 3] | 0.03 [0 to 1]

3. Secondary Outcome: Number of Participants With Malpositions
Time Frame: Measured from initiation to completion of procedure (usually from 0 to 300 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (Chest X-ray) | Sherlock 3CG® TCS
Number analyzed (Participants) | 60 | 60
Participants | 12 | 0

4. Secondary Outcome: Number of Subsequent Malposition Attempts
Description: This is the number of remaining malpositions following the first malposition adjustment attempt. All PICCs were inserted properly after the second malposition adjustment attempt.
Time Frame: Measured from initiation to completion of procedure (usually from 0 to 300 minutes)
Measure: Number; unit: malposition adjustment attempts
Arm/Group | Standard of Care (Chest X-ray) | Sherlock 3CG® TCS
Number analyzed (Participants) | 60 | 60
malposition adjustment attempts | 12 | 0

5. Secondary Outcome: Health Care Professional (HCP) Procedural Satisfaction (Overall)
Description: HCPs were asked to rate satisfaction with the procedure (overall) on a scale from 0 to 10 with 0 meaning "not at all satisfied" and 10 meaning "extremely satisfied".
Time Frame: Measured immediately after the procedure completion (usually ranges from 0 to 300 minutes following procedure initiation).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (Chest X-ray) | Sherlock 3CG® TCS
Number analyzed (Participants) | 60 | 60
units on a scale | 6.22 (2.90) | 9.22 (1.55)

6. Secondary Outcome: Number of Additional Venous Access Devices (VADs) Required Due to PICC Not Being Ready for Use
Time Frame: Measured from initiation to completion of procedure (usually from 0 to 300 minutes)
Measure: Number; unit: Venous Access Devices (VADs)
Arm/Group | Standard of Care (Chest X-ray) | Sherlock 3CG® TCS
Number analyzed (Participants) | 60 | 60
Venous Access Devices (VADs) | 0 | 0

7. Secondary Outcome: Number of Medication Doses Missed Due to PICC Not Being Ready for Use
Time Frame: Measured from initiation to completion of procedure (usually from 0 to 300 minutes)
Measure: Mean (Standard Deviation); unit: Doses
Arm/Group | Standard of Care (Chest X-ray) | Sherlock 3CG® TCS
Number analyzed (Participants) | 60 | 60
Doses | 0.07 (0.31) | 0 (0)

8. Secondary Outcome: Number of Lab Draws Missed Due to PICC Not Being Ready for Use
Time Frame: Measured from initiation to completion of procedure (usually from 0 to 300 minutes)
Measure: Mean (Standard Deviation); unit: Lab draws
Arm/Group | Standard of Care (Chest X-ray) | Sherlock 3CG® TCS
Number analyzed (Participants) | 60 | 60
Lab draws | 0.07 (0.25) | 0 (0)

9. Secondary Outcome: Number of Overtime Hours Worked Per PICC Placement Procedure
Time Frame: Measured from initiation to completion of procedure (usually from 0 to 5 hours)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Standard of Care (Chest X-ray) | Sherlock 3CG® TCS
Number analyzed (Participants) | 60 | 60
hours | 0.07 (0.25) | 0 (0)

10. Other Pre Specified Outcome: Nurse Time Associated With Initial PICC Placement (Per Patient)
Description: Nurse time associated with initial PICC placement was defined as the time between when the nurse arrived at the subject and when the nurse left the room, minus the amount of time it took to conduct the research consent with the subject for the study; it includes time spent gathering supplies (before entering the subject's room) and any consents obtained for the PICC procedure (not study-related consents).
Time Frame: Usually ranges from 0 to 150 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Standard of Care (Chest X-ray) | Sherlock 3CG® TCS
Number analyzed (Participants) | 60 | 60
minutes | 42.50 (16.81) | 42 (16.35)

11. Other Pre Specified Outcome: Nurse Time Associated With Malposition Adjustment After Initial PICC Placement (Per Event)
Description: Nurse time associated with a malposition was defined as the time between when the nurse opened gathered materials for correcting the malposition (e.g., PICC kit, dressing change kit, saline, syringe) and when the subject was released for IV therapy.
Time Frame: Usually ranges from 0 to 30 minutes
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: events
Arm/Group | Standard of Care (Chest X-ray)
Number analyzed (Participants) | 7
Number analyzed (events) | 7
minutes | 11.67 (10.5)

12. Other Pre Specified Outcome: Mean Total Procedural Cost From Initiation of Procedure (Opening of PICC Kit) to Catheter Tip Confirmation (Release for IV Therapy)
Description: Cost calculated as follows: mean (sum of material cost per PICC insertion, X-ray cost per PICC insertion, non-interventional radiology (IR) labor cost per PICC insertion, IR labor cost per PICC insertion).
Time Frame: Usually ranges from 0 to 300 minutes
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | Standard of Care (Chest X-ray) | Sherlock 3CG® TCS
Number analyzed (Participants) | 60 | 60
US dollars | 367 (324.21) | 272 (67.03)

ADVERSE EVENTS:
Time Frame: Subjects were followed only up to the point at which the PICC line tip was confirmed and they were released to receive therapy (usually from 0 to 300 minutes following procedure initiation). Once they were released to receive therapy, and review of electronic medical record (EMR) data was complete, there was no other subject follow-up.
Arm/Group | Standard of Care (Chest X-ray) | Sherlock 3CG® TCS
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No